CLINICAL TRIAL: NCT02383251
Title: A Randomized Phase II Study of Pazopanib and Weekly Paclitaxel in Patients With Platinum Resistant/Refractory Ovarian Cancer Who Relapse During Bevacizumab Maintenance
Brief Title: Paclitaxel/Pazopanib for Platinum Resistant/Refractory Ovarian Cancer
Acronym: TAPAZ
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-OV231
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — pazopanib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pazopanib/Paclitaxel association (Experimental): Arm 1 :
  Pazopanib alone during 1 week at 600 mg (1x400mg and 1x200mg), per day, taken orally without food at least one hour before or two hours after a meal.
  Then:
  * Pazopanib 600 mg (1x400mg and 1x200mg), per day, taken orally without food at least one hour before or two hours after a meal.
  * Paclitaxel 65 mg/m2 i.v. on days 1, 8, 15 every 28 days until progression of disease or toxicity
  Interventions: Drug: Pazopanib; Drug: Paclitaxel
- Paclitaxel alone (Active Comparator): Arm 2 :
  * Paclitaxel 80mg/m2 i.v. on days 1, 8, 15
  * every 28 days until progression of disease or toxicity
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Pazopanib — Pazopanib 600mg during the fist cycle. Then, if there is not heptic triuyble, the dose could be increased to 800mg
  Other Names: Votrient
  Arms: Pazopanib/Paclitaxel association
Drug: Paclitaxel — Arm 1 : Paclitaxel 65mg/m² Arm 2: Paclitaxel 80mg/m²
  Other Names: Taxol

SUMMARY:
Study of Pazopanib and weekly Paclitaxel in patients with platinum resistant/refractory ovarian cancer who relapse during bevacizumab maintenance.

DETAILED DESCRIPTION:
Standard of treatments:

* In Europe, advanced ovarian cancer patients are treated in first line with optimal debulking surgery followed by carboplatin/paclitaxel regimen plus bevacizumab during chemotherapy and as maintenance for a total à 15 months. The addition of bevacizumab is a standard for the patients with residual disease.
* The addition of bevacizumab to carboplatin/gemcitabine chemotherapy was also recently approved for patients with platinum sensible relapse [Aghajanian, 2012]. The bevacizumab is maintained until progression.

Rationale to use anti-angiogenic agents in early relapse:

* The recent AURELIA trial comparing paclitaxel, topotecan or liposomal doxorubicin alone versus combined to bevacizumab after early failure of the first-line with carboplatin/paclitaxel revealed that targeting angiogenesis was beneficial in recurrent platinum-resistant ovarian cancer [Pujade-Lauraine, 2012 and 2013], with higher progression-free survival (PFS). Thus, the strategy of inhibiting angiogenesis in recurrent resistant-platinum ovarian cancer is very promising.
* The recent changes of the standard of treatment of first line and platinum-sensible relapse of patients with ovarian cancer highlights the question of inhibiting angiogenesis for relapse during/after bevacizumab maintenance. In this last situation, the strategy of continuation of antiangiogenesis therapy, just in changing chemotherapy despite recurrence, showed benefit in other types of cancer (colon, lung). In ovarian cancer, no study has been performed to answer to the question. In Aurelia trial, However, patients did not previously receive bevacizumab.

The choice of the best antiangiogenic agent in alternative to bevacizumab needs to be assessed. Small molecular inhibitor of tyrosine-protein-kinases (TK) could be used with efficacy after a first-line of antiangiogenesis treatment as it was demonstrated in renal cancer [Escudier, 2011].

* Pazopanib is an oral, potent multi-targeted small-molecule inhibitor of VEGF-receptor TKs (VEGFR-1 -2 -3 PDGFR and c-KIT; it is the first targeted small molecule that it has demonstrated an important activity in ovarian cancer. At ASCO 2013, the AGO-OVAR16 trial of maintenance of pazopanib in first line ovarian cancer has shown a benefit in progression free survival (difference of 5.6 months of median PFS in favour of pazopanib compared to placebo) [Dubois, ASCO 2013 LBA5503]; in this trial, the majority of the patients had few residual disease and patients did not receive bevacizumab.
* In ovarian cancer, the standard treatment for patients relapsing during bevacizumab maintenance (15 to 20% of patients) is still a mono-chemotherapy. Weekly paclitaxel is one oh the most commonly used chemotherapy in this situation of early relapse. However, the promising results of pazopanib in first line led to develop protocols in second-line in combination with chemotherapy.

The combination of weekly paclitaxel and pazopanib is feasible and the dose proposed for further phase 2 studies is pazopanib 800 mg daily and paclitaxel 65 mg/m2 at day 1, 8, 15 every 28 days [Tan, the oncologist 2010]. The dosage of paclitaxel was justified on results from previous studies, demonstrating that co-administration of pazopanib and paclitaxel increases the systemic exposure to paclitaxel. An Italian group has just closed a phase 2 study (MITO11) that evaluated this association among ovarian patients with early relapse. In this study, patients did not receive previously bevacizumab.

Thus, pazopanib is the best molecule to be associated to chemotherapy in ovarian cancer patients who early relapse after a treatment including bevacizumab.

We propose a randomized phase 2 trial to evaluate the combination of pazopanib to weekly paclitaxel among patients with platine resistant relapse after treatment including bevacizumab maintenance

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Performance status ECOG < 2
3. Histological documented ovarian, tubal or peritoneum carcinoma (stage IC to IV)
4. Patient treated at least with one line of platinum-based chemotherapy who have relapsed within 6 months after trhe last administration of platinum-based chemotherapy and taking bevacizumab for maintenance NB: Penultimate line of chemotherapy could contain chemotherapy without platinum and the last line should contain platinum-based chemotherapy (followed by bevacizumab for maintenance)
5. Patients must have disease that is measurable and/or evaluable according to RECIST criteria and requires chemotherapy treatment
6. Patients with liver metastasis can be included
7. Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow up.
8. Life expectancy of more than 3 months
9. Able to swallow and retain oral medication
10. Adequate organ system function like:

Total bilirubin ≤ 1.5 X ULN Alanine amino transferase (ALT) and Aspartate aminotransferase (AST)c ≤ 2.5 X ULN

1. Subjects may not have had a transfusion within 7 days of screening assessment.
2. Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.
3. Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN (upper limit of normal) are not permitted.
4. If UPC <1, then a 24-hour urine protein must be assessed. Subjects must have a 24-hour urine protein value <1 g to be eligible. Use of urine dipstick for renal function assessment is not acceptable. 10. Women of childbearing potential must agree to use effective contraception 11. Negative serum pregnancy test (if applicable) 12. Affiliated to or a beneficiary of a social security category

Exclusion Criteria:

1. Prior malignancy over the past 5 years with the exception of in situ carcinomas of the cervix or basal and squamous cell carcinoma or nonmelanoma skin cancer properly treated, or all solid tumor, considered as in completed remission without relapse for at least 5 years
2. Central nervous system (CNS) metastases at baseline, with the exception of those subjects who have previously-treated CNS metastases (surgery ± radiotherapy) and who meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or enzyme-inducing anticonvulsants of P3A4 cytochrom
3. Previous treatment with monotherapy weekly paclitaxel
4. Previous treatment with bevacizumab within three weeks before start of studt treatment
5. Patients with severe hypersensitivity to a product containing castor oil polyoxyl 35 or paclitaxel solvent: the Chremophor
6. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

   * Active peptic ulcer disease
   * Known intraluminal metastatic lesion/s with risk of bleeding
   * Inflammatory bowel disease (e.g. ulcerative colitis, Chrohn's disease), or other gastrointestinal conditions with increased risk of perforation
   * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
7. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

   * Malabsorption syndrome
   * Major resection of the stomach or small bowel.
8. Corrected QT interval (QTc) > 450 msecs or > 480 msecs for patient with block branch
9. History of any one or more of the following cardiovascular conditions within the past 6 months:

   * Cardiac angioplasty or stenting
   * Myocardial infarction
   * Unstable angina
   * Coronary artery bypass graft surgery
   * Symptomatic peripheral vascular disease
   * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
   * Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].
10. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible
11. Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major surgery).
12. to 14: All risk of bleeding

15 Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures. 16 Unable or unwilling to discontinue use of prohibited medications 17 Treatment with any of the following anti-cancer therapies:

* radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib (out of bevacizumab) OR
* chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of pazopanib (out of bevacizumab) 18 Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment 19 Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia. 20 Patient deprived of liberty or state-controlled 21 Inability to participate to medical follow up for geographic

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 4 months
  Proportion of progression or death 4 months after initiation of treatment

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  Time between randomization and death or last news date for patient alive at the last visit date
Disease control rate (DCR) | Up to 2 years
  Proportion of woman in partial, compete or stable desease according to RECIST 1.1. criteria
Toxicity according to NCI CTCAE v4.3 criteria | Up to 2 years
  tolerance of the treatment based on AE occurrence according to NCI CTCAE v4.3 criteria
health-related quality of life | Up to 2 years
  health-related quality of life and symptomatic state will be evaluated by filing questionnaires by patients

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY, PHD, Principal Investigator — Centre François Baclesse, Caen
Locations (36):
- France (36):
  - Hôpital Henri Duffaut, Avignon
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier de Dax, Dax
  - Centre Georges François Leclerc, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Hôpital Michallon - Centre Hospitalier Universitaire de Grenoble, Grenoble
  - Hôpital André Mignot, Le Chesnay
  - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - Hôpital de la Croix Rousse, Lyon
  - Centre Léon Bérard, Lyon
  - Hôpital Européen, Marseille
  - Institut Paoli Calmettes, Marseille
  - Hôpital de Mont-de-Marsan, Mont-de-Marsan
  - ICM Val d'Aurelle, Montpellier
  - ORACLE - Centre d'Oncologie de Gentilly, Nancy
  - Centre Catherine de Sienne, Nantes
  - Centre ONCOGARD - Institut de Cancérologie du Gard, Nîmes
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Université Paris Descartes, AP-HP, Hôpitaux Universitaires Paris Centre, Site Cochin, Paris
  - Clinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - HPCA - Hôpital Privé des Côtes d'Armor, Plerin SUR MER
  - "Hôpital de la Milétrie - Centre Hospitalier Universitaire de Poitiers - Pôle Régional de Cancérologie", Poitiers
  - Institut du Cancer Courlancy Reims, Reims
  - ICO Centre René Gauducheau, Saint-Herblain
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Centre Paul Strauss, Strasbourg
  - Centre Hospitalier de Thonon-les-Bains, Thonon-les-Bains
  - Centre Hospitalier Universitaire Bretonneau, Tours
  - ICL Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Joly F, Fabbro M, Berton D, Lequesne J, Anota A, Puszkiel A, Floquet A, Vegas H, Bourgeois H, Bengrine Lefevre L, You B, Pommeret F, Lortholary A, Spaeth D, Hardy-Bessard AC, Abdeddaim C, Kaminsky-Forrett MC, Tod M, Kurtz JE, Del Piano F, Meunier J, Raban N, Alexandre J, Mouret-Reynier MA, Ray-Coquard I, Provansal Gross M, Brachet PE. Paclitaxel with or without pazopanib for ovarian cancer relapsing during bevacizumab maintenance therapy: The GINECO randomized phase II TAPAZ study. Gynecol Oncol. 2022 Sep;166(3):389-396. doi: 10.1016/j.ygyno.2022.06.022. Epub 2022 Jul 26. PMID 35902297